CLINICAL TRIAL: NCT06081036
Title: Courbes Normatives De Volumes Cérébraux Issues D'IRM Fœtales Multicentriques
Brief Title: Normative Brain Volume Profiles From Multicenter Fetal MRI
Acronym: MULTINORMFET
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0324
Record Dates: First submitted 2023-05-25; First posted 2023-10-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cortical Development Malformation; Multiparametric Magnetic Resonnance Imaging; Brain Cortical Thickness; Prenatal Diagnosis; Fetal Development
MeSH Terms: conditions — Malformations of Cortical Development | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire about children development

SUMMARY:
Fetal brain MRI is an essential diagnostic tool to inform parents about the prognosis of abnormalities detected on routine ultrasound. Recent work has shown that brain MRI measurements at the antenatal stage are predictive of the child's postnatal development. However, this work remains limited to basic research, in part because of the lack of normative curves of brain tissue volume evolution from fetal MRI acquired in clinical routine. This project aims to fill this gap. For this purpose, the project will exploit fetal MRI scans acquired in 4 French hospitals (Marseille, Nice, Montpellier and Paris): MRI scans without abnormalities will be centralized for analysis, and families who have undergone these scans will be contacted to evaluate the development of their children after birth. Normative curves will be established by applying a set of treatments developed by the laboratory in Marseille collaborating in the project. Ultimately, these curves will help to clarify the diagnosis of fetuses by providing a quantitative characterization of the normality of brain measurements.

ELIGIBILITY:
Inclusion Criteria:

Child who has had, more than 3 years ago, a cerebral MRI during the fetal period in one of the 4 partner centers

Exclusion Criteria:

* Child suffering from a commissural malformation (anomaly of the corpus callosum)
* Child with a genetic syndrome and/or chromosomal abnormality and/or deleterious mutation
* Child with syndromic extra-cerebral malformations (including cardiac malformations)
* Child with intrauterine growth restriction reported in the obstetrical record
* Child with maternal-fetal infection (TORCH, parvovirus or other) confirmed by amniotic fluid test or neonatal urine test
* Multiple pregnancy
* Mother with diabetes treated during pregnancy (including gestational diabetes, if treated)
* Mother with antiepileptic medication during pregnancy
* Alcohol or drug use
* Presence of a sustentorial arachnoid cyst
* Presence of an arachnoid cyst with mass effect
* Objection from parental authority holders to participate in the study

Ages: 20 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Homogeneous group of fetuses who received an MRI more than 3 years ago, with normal MRI and normal neurological development at 3 years (see inclusion criteria). Included individuals (at the fetal stage) will be evaluated at 3+ years post-birth.
Sampling Method: Non-Probability Sample
Enrollment: 1423 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine normative brain volume curves | Through study completion, an average of 3 year
  Curves calculated from fetal brain MRIs in fetuses between 20 and 37 weeks of amenorrhea with normal postnatal neurological development

SECONDARY OUTCOMES:
Statistically compare the normative curves obtained with standard articles in the literature. | Through study completion, an average of 3 year
  Comparaison of Size effect, confidence intervals obtained with those reported in the reference articles
Sensitivity study: Possible influence of the scanner type on the estimated normative curves. | Through study completion, an average of 3 year
  MRI scanner model

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No